CLINICAL TRIAL: NCT00922922
Title: Duration and Direct Cost of Behavioral Health Concerns in Pediatric Primary Care
Acronym: EI
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0136-09-EP
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the duration and direct cost of pediatric primary care visits consisting of medical concerns only, behavioral concerns only, and medical and behavioral concerns.

DETAILED DESCRIPTION:
Behavioral, emotional, and psychosocial issues of children and adolescents are often brought to the attention of primary care physicians by parents (Smith, Rost, & Kashner, 1995). In fact, behavioral health concerns are the primary reason for visits to physicians in 15% to 21% of cases (Kelleher, Childs, Wasserman, McInerny, Nutting, & Gardner, 1997; Lavigne, Gibbons, Arend, Rosenbaum, Binns, & Christoffel, 1999; Williams, Klinepeter, Palmes, Pulley, & Foy, 2004). During 50% to 80% of child health care visits, parents or physicians raise concerns of behavioral or psychosocial issues (Cassidy & Jellinek 1998; Fries, Koop, Beadle, Cooper, England, Greaves, et al., 1993; Sharp, Pantell, Murphy, & Lewis, 1992).

Several concerns have been raised when patients seek mental health services from primary care physicians, including an increase in the number of medical visits, an increase in the time spent with the physician, lost revenue if a patient takes more time than scheduled, a lower reimbursement rate for mental health issues, limited training in mental health treatment, a decrease in the number of patients seen, an increase in the risk of physician burnout, unsatisfied patients, an increase in impairment in patient health and functioning, and an increase in the use of acute and emergency care (Connor, McLaughlin, Jeffers-Terry, O'Brien, Stille, Young, & Antonelli, 2006; deGruy, 1997; Leaf, Owens, Levelthal, Forsyth, Vaden-Kiernan, Epstein, et al., 2004; Strosahl, 2002; Young, Klap, Sherbourne, & Wells, 2001).

There are limited studies examining the time and cost incurred by physicians for treating patients with behavioral, emotional, and psychosocial issues. Average primary care visits last between 13 and 17 minutes (Blumenthal, Causino, Chang, Culpepper, Marder, Saglam, et al., 1999; Bryant & Shimizu, 1988) A more recent study conducted in rural communities found that physicians spent an average of 5 to 7 minutes longer on visits where behavioral issues were raised (Cooper, Valleley, Polaha, Begeny, & Evans, 2006). Primary care physicians see four or five patients per hour (deGruy, 1997), which is an insufficient amount of time for a detailed psychological assessment or management of mental health symptoms. Therefore, frequent or longer visits are scheduled. Additionally, physicians are reimbursed for medical diagnosis but not mental diagnoses (deGruy).

This study is based on previous work documenting that pediatric primary care visits increased in duration when behavioral concerns were identified prior to the visit and spontaneously raised during the visit (Cooper, et al., 2006). Additionally, this study calculates the reimbursement rate associated with those visits in addition to the duration of the visit. Finally, this study is a replication of a study previously approved through the University of Nebraska Medical Center Institutional Review Board (i.e., IRB # 449-07-EP).

ELIGIBILITY:
Inclusion Criteria:

* Patients who attend a local pediatrician clinic between between March 2009 and March 2010

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 500 patients from a pediatrician office will be reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2009-04-03 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Valleley, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Munroe Meyer Institute, Omaha, Nebraska, United States